CLINICAL TRIAL: NCT02395770
Title: Effects of a Movement Training Oriented Rehabilitation Program on Symptoms, Functional Limitations and Acromiohumeral Distance in Individuals With Subacromial Pain Syndrome
Brief Title: Effects of a Movement Training for Subacromial Pain Syndrome
Acronym: MTforSPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OPPQ-Apr2013
Record Dates: First submitted 2015-03-09; First posted 2015-03-24 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Shoulder Impingement Syndrome
Keywords: Shoulder; Rotator cuff; Rehabilitation; Motor control
MeSH Terms: conditions — Shoulder Impingement Syndrome | interventions — Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Subacromial pain group (Experimental): Rehabilitation Program: The program was developed to target the deficits described in individuals with SPS. It included movement training, manual therapy, strengthening and stretching exercises, and patient education. Each supervised session lasted around 30 minutes, with 75% of the session for movement training. Three treating physiotherapists supervised the program and initially attended a training session to standardize the program.
  Interventions: Other: Rehabilitation program

INTERVENTIONS:
Other: Rehabilitation program — Movement training: To re-educate control of movement, exercises of increasing difficulty in terms of movement plane, range of motion, speed and resistance were performed.
  Strengthening: Using extremities weight, free weights or elastic bands, scapulothoracic and scapulohumeral strengthening was performed to increase strength and control of shoulder muscles.
  Stretching & Manual Therapy: These modalities, performed only if needed, were aimed at addressing stiffness of posterior and inferior glenohumeral capsule and pectoralis minor.
  Patient education: Participants received education regarding posture and body mechanics. They were instructed on preferred shoulder positioning during sleep, activities, work and sports

SUMMARY:
Objectives: Evaluate the effects of a rehabilitation program based on movement training on symptoms, functional limitations and acromiohumeral distance (AHD) in individuals with SPS.

Methods: Twenty-five participants with SPS participated in a 6-week program. Outcomes of both groups were evaluated at baseline and 6 weeks. Changes in symptoms and functional limitations were assessed. Changes in AHD for both groups were assessed using ultrasonographic measures.

DETAILED DESCRIPTION:
Background: Multiple factors have been associated with the presence of a subacromial pain syndrome (SPS), including deficits in performance of scapular and glenohumeral muscles. Such deficits can lead to inadequate kinematics and decreased acromiohumeral distance (AHD). Exercises that aim at correcting these deficits, such as movement training, were suggested to improve symptoms and functional limitations. To date, few studies have assessed outcomes following an intervention focused on movement training.

Objectives: Evaluate the effects of a rehabilitation program based on movement training on symptoms, functional limitations and AHD in individuals with SPS.

Design: Prospective single group pre-post design. Methods: Twenty-five participants with SPS (SPS group) participated in a 6-week program. Twenty asymptomatic volunteers were recruited for normative AHD values (control group). Outcomes of both groups were evaluated at baseline and 6 weeks, i.e. immediately following intervention for the SPS group. Changes in symptoms and functional limitations for SPS group were assessed using the Western Ontario Rotator Cuff index (WORC) and Disability of the Arm Shoulder and Hand questionnaire (DASH). Changes in AHD for both groups were assessed using ultrasonographic measures.

ELIGIBILITY:
Inclusion Criteria:

* painful arc of movement during flexion or abduction
* positive Neer or Kennedy-Hawkins impingement signs
* pain on resisted lateral rotation, abduction or empty can test.

Exclusion Criteria:

* previous shoulder surgery
* shoulder pain reproduced by neck movement
* clinical signs of full-thickness RC tears
* shoulder capsulitis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2013-06; Primary Completion 2014-05 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Symptoms and functional limitations - Upper limb | week 6
  Upper limb symptoms and functional limitations were assessed using the Disability of the Arm Shoulder and Hand (DASH) questionnaire. DASH has 30 items that measures upper limb physical disability and symptoms. Final scores range from 0 to 100 (most severe disability).

SECONDARY OUTCOMES:
Symptoms and functional limitations - Shoulder | week 6
  Shoulder symptoms and functional limitations was assessed using the Western Ontario Rotator Cuff (WORC) index. The WORC is a disease-specific questionnaire designed for patients with RC disorders. Scores vary from 0 to 100 (high functional status).
Ultrasonographic measurements of acromiohumeral distance (AHD) | week 6
  Measurement of AHD is defined as the tangential distance between the bony landmarks of humeral head and inferior edge of acromion, corresponding to the anterior outlet of subacromial space.Measurements were taken in a sitting position with the arm at rest, and at 45° and 60° of active abduction.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Sébastien Roy, PhD, Principal Investigator — Centre interdisciplinaire de recherche en réadaptation et en intégration sociale (CIRRIS)
Locations (1):
- Centre for Interdisciplinary Research in Rehabilitation and Social Integration, Québec, Quebec, Canada

REFERENCES:
- [Background] Desmeules F, Minville L, Riederer B, Cote CH, Fremont P. Acromio-humeral distance variation measured by ultrasonography and its association with the outcome of rehabilitation for shoulder impingement syndrome. Clin J Sport Med. 2004 Jul;14(4):197-205. doi: 10.1097/00042752-200407000-00002. PMID 15273525
- [Background] Ngomo S, Mercier C, Bouyer LJ, Savoie A, Roy JS. Alterations in central motor representation increase over time in individuals with rotator cuff tendinopathy. Clin Neurophysiol. 2015 Feb;126(2):365-71. doi: 10.1016/j.clinph.2014.05.035. Epub 2014 Jun 21. PMID 25043198
- [Background] Roy JS, Moffet H, McFadyen BJ. The effects of unsupervised movement training with visual feedback on upper limb kinematic in persons with shoulder impingement syndrome. J Electromyogr Kinesiol. 2010 Oct;20(5):939-46. doi: 10.1016/j.jelekin.2009.10.005. Epub 2009 Nov 8. PMID 19900823
- [Background] Roy JS, Moffet H, Hebert LJ, Lirette R. Effect of motor control and strengthening exercises on shoulder function in persons with impingement syndrome: a single-subject study design. Man Ther. 2009 Apr;14(2):180-8. doi: 10.1016/j.math.2008.01.010. Epub 2008 Mar 20. PMID 18358760
- [Derived] Savoie A, Mercier C, Desmeules F, Fremont P, Roy JS. Effects of a movement training oriented rehabilitation program on symptoms, functional limitations and acromiohumeral distance in individuals with subacromial pain syndrome. Man Ther. 2015 Oct;20(5):703-8. doi: 10.1016/j.math.2015.04.004. Epub 2015 Apr 14. PMID 25907145